CLINICAL TRIAL: NCT02110082
Title: A Phase 1b, Open-label, Multicenter Study of Urelumab (BMS-663513) in Combination With Cetuximab in Subjects With Advanced/Metastatic Colorectal Cancer or Advanced/Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Combination Study of Urelumab and Cetuximab in Patients With Advanced/Metastatic Colorectal Cancer or Advanced/Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA186-018
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer; Head and Neck Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms | interventions — urelumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Urelumab + Cetuximab (Experimental): Urelumab every 3 weeks with Cetuximab weekly through Intravenous infusion
  Interventions: Biological: Urelumab; Biological: Cetuximab
- Cohort 2: Urelumab + Cetuximab (Experimental): Urelumab every 3 weeks with Cetuximab weekly through Intravenous infusion
  Interventions: Biological: Urelumab; Biological: Cetuximab

INTERVENTIONS:
Biological: Urelumab
  Other Names: BMS-663513
Biological: Cetuximab

SUMMARY:
The purpose of the study is to determine the safety, tolerability and maximum tolerated dose of Urelumab in combination with Cetuximab in patients with Advanced/Metastatic Colorectal Cancer or Advanced/Metastatic Squamous Cell Carcinoma of the Head and Neck.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects with advanced/metastatic Colorectal Cancer(CRC) who have failed or been intolerant to both irinotecan- and oxaliplatin- based regimens
* Subjects with advanced/metastatic Squamous cell carcinoma of the head and neck (SCCHN) who are without options for curative treatment
* Subjects must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Men and women 18 and older
* Women of childbearing potential (WOCBP) and men must use highly effective methods of contraception
* Eastern Cooperative Oncology Group (ECOG) of 0 or 1
* Subjects must have a life expectancy of at least 3 months

Exclusion Criteria:

* Active or progressing brain metastases
* Other concomitant malignancies (with some exceptions per protocol)
* Nasopharyngeal carcinoma
* Active or history of autoimmune disease
* Positive test for Human Immunodeficiency Virus (HIV) 1&2 or known AIDS
* History of any hepatitis (A,B or C)
* Known current drug or alcohol abuse
* Active Tuberculosis (TB)
* Use of anti-cancer treatments within 28 days
* Prior therapy with anti-CD137 antibody

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint is the incidence, potential significance, and clinical importance of adverse events | Approximately 2 years
  As determined by medical review of adverse event reports, vital sign measurements, electrocardiograms (ECGs), and results of physical examination and laboratory tests During a 3 week cycle, safety labs are done on Days 1, 2, 3, 5, 8, and 15. Starting on Cycle 3, Day 1, Chemistry (excluding Liver function test (LFTs)) are to be performed on Day 1 and Day 15 of each cycle thereafter. Physical exams are done on Day 1 of each cycle. Vital signs are done on Days 1, 2, 8, and 15 at Cycle 1 and then on Days 1 and 2 of each cycle thereafter. Adverse events are collected from screening to 60 days after last dose of Urelumab

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
Duration of Objective Response (DOR) | Up to 2 years
Progression Free Survival (PFS) | Up to 2 years
Immunogenicity measured by the occurrence of anti-drug antibody after the administration of BMS-663513 | Up to 2 years
Maximum observed serum concentration (Cmax) of BMS-663513 in combination with Cetuximab | Up to 2 years
Time of maximum observed serum concentration (Tmax) of BMS-663513 in combination with Cetuximab | Up to 2 years
Area under the serum concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of BMS-663513 in combination with Cetuximab | Up to 2 years
Area under the serum concentration-time curve from time zero to the time of last quantifiable serum concentration (AUC(0-T)) of BMS-663513 in combination with Cetuximab | Up to 2 years
Elimination half-life (T-HALF) of BMS-663513 in combination with Cetuximab | Up to 2 years
Total body clearance (CLT) of BMS-663513 in combination with Cetuximab | Up to 2 years
Volume of distribution at steady-state (Vss) of BMS-663513 in combination with Cetuximab | Up to 2 years
Trough observed concentration (Cmin) of BMS-663513 in combination with Cetuximab | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (7):
  - Stanford University, Stanford, California
  - University Of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Providence Oncology & Hematology Care Eastside, Portland, Oregon
  - Upmc Cancer Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Khushalani NI, Ott PA, Ferris RL, Cascone T, Schadendorf D, Le DT, Sharma MR, Barlesi F, Sharfman W, Luke JJ, Melero I, Lathers D, Neely J, Suryawanshi S, Sanyal A, Holloway JL, Suryawanshi R, Ely S, Segal NH. Final results of urelumab, an anti-CD137 agonist monoclonal antibody, in combination with cetuximab or nivolumab in patients with advanced solid tumors. J Immunother Cancer. 2024 Mar 7;12(3):e007364. doi: 10.1136/jitc-2023-007364. PMID 38458639
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx